CLINICAL TRIAL: NCT06714422
Title: Should Doctors Bring an Apple to Have a More Relaxed Night Shift?: a Single Center, Open Label, Randomized Trial
Brief Title: Apples in Night Shift
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Li Rong, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APPLE study
Record Dates: First submitted 2024-11-21; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Night Work
Keywords: night shift; apple; doctor; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- no apple group (Active Comparator): No apples during night shift
  Interventions: Procedure: no apple group
- apple group (Experimental): Doctors will bring apples during night shift
  Interventions: Procedure: apple group

INTERVENTIONS:
Procedure: apple group — Doctors will bring apples during night shift
  Arms: apple group
Procedure: no apple group — No apples during night shift
  Arms: no apple group

SUMMARY:
Background: Emergency doctors face a highly stressful work environment during night shifts. Long-term night shift work can lead to sleep deprivation, fatigue accumulation, and disruption of the biological clock, which may affect doctors' work efficiency and physical and mental health. There are various health interventions for night shift doctors, one of which is an interesting practice of carrying an apple as a symbol of the "night shift deity" to relieve anxiety and improve work efficiency. Although this behavior is not supported by sufficient scientific evidence, it has become a common habit among some doctors during night shifts due to its simplicity, low risk, and ritualistic nature.

Objective: To assess whether carrying an apple during night shifts can significantly reduce fatigue, decrease work intensity, and enhance work experience for emergency doctors.

Design: Single-center, open-label, randomized controlled trial.

Participants: several doctors with a total of 60 emergency working night shifts.

Primary Outcome: Average number of patients per night shift.

Sample Size: The study plans to recruit several doctors with a total of 60 emergency night shifts and randomly assign them to the experimental group and the control group. One doctor can be randomized for many times.

DETAILED DESCRIPTION:
Background: Emergency doctors face a highly stressful work environment during night shifts. Long-term night shift work can lead to sleep deprivation, fatigue accumulation, and disruption of the biological clock, which may affect doctors' work efficiency and physical and mental health. There are various health interventions for night shift doctors, one of which is an interesting practice of carrying an apple as a symbol of the "night shift deity" to relieve anxiety and improve work efficiency. Although this behavior is not supported by sufficient scientific evidence, it has become a common habit among some doctors during night shifts due to its simplicity, low risk, and ritualistic nature.

Objective: To assess whether carrying an apple during night shifts can significantly reduce fatigue, decrease work intensity, and enhance work experience for emergency doctors.

Design: Single-center, open-label, randomized controlled trial.

Participants: several doctors with a total of 60 emergency working night shifts.

Primary Outcome: Average number of patients per night shift.

Sample Size: The study plans to recruit several doctors with a total of 60 emergency night shifts and randomly assign them to the experimental group and the control group. One doctor can be randomized for many times.

ELIGIBILITY:
Inclusion Criteria:

Doctors who have a night shift in the emergency department of gynaecology with at least two weeks experience.

Exclusion Criteria:

Doctors who refuse to join the study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
number of patients | from 5pm on the Randomization day to 8am on the next day
  Number of patients during the night shift

SECONDARY OUTCOMES:
Evaluation of night shifts | from 5pm on the Randomization day to 8am on the next day
  Overall evaluation of night shifts by doctors (Good, Average, Poor)
Emergency admissions | from 5pm on the Randomization day to 8am on the next day
  Admissions of emergency patients during the night shift randomized.
Emergency surgery number | from 5pm on the Randomization day to 8am on the next day
  Number of patients who experience emergency surgery during the night shift.
Emergency uterine evacuation number | from 5pm on the Randomization day to 8am on the next day
  Number of patients who need emergency uterine evacuation during the night shift.
Complicated patients number | from 5pm on the Randomization day to 8am on the next day
  The number of patients needs to be checked by a senior doctor
Doctor's break time | from 5pm on the Randomization day to 8am on the next day
  The time (hours) of the doctor's break.
Number of patients admitted to emergency room | from 5pm on the Randomization day to 8am on the next day
  The number of people who need to be admitted to the emergency room

IPD SHARING:
Plan to Share IPD: Yes
all night shift data
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available when they have been published in journals.
Access Criteria: Please contact investigator Kai-Lun Hu. hukailun@bjmu.edu.cn